CLINICAL TRIAL: NCT00074269
Title: Pilot Study Of Allogeneic Peripheral Blood Progenitor Cell Transplantation In Patients With Chemotherapy-Refractory Or Poor-Prognosis Metastatic Breast Cancer
Brief Title: Allogeneic Stem Cell Transplant After ATG, High-Dose Melphalan, and Fludarabine for Patients With Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to poor enrollment
Sponsor: University of California, San Diego (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Edward Ball, MD, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020815; CDR0000343758 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Antilymphocyte Serum; Filgrastim; Cyclosporine; fludarabine phosphate; Melphalan; Methotrexate; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment (Experimental)
  Interventions: Biological: anti-thymocyte globulin; Biological: filgrastim; Biological: graft-versus-tumor induction therapy; Biological: therapeutic allogeneic lymphocytes; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: melphalan; Drug: methotrexate; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin
Biological: filgrastim
Biological: graft-versus-tumor induction therapy
Biological: therapeutic allogeneic lymphocytes
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: melphalan
Drug: methotrexate
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving chemotherapy, such as fludarabine and melphalan, before a donor peripheral blood stem cell transplant helps stop the growth of tumor cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining tumor cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells (donor lymphocyte infusion) after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving antithymocyte globulin, cyclosporine, and methotrexate before or after the transplant may stop this from happening.

PURPOSE: This phase II trial is studying how well antithymocyte globulin, high-dose melphalan, fludarabine, and allogeneic peripheral stem cell transplant work in treating patients with metastatic adenocarcinoma of the breast.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity and tolerability of allogeneic peripheral blood stem cell transplantation after a nonmyeloablative preparative regimen comprising anti-thymocyte globulin, high-dose melphalan, and fludarabine in women with chemotherapy-refractory or poor-prognosis metastatic adenocarcinoma of the breast.
* Determine the ability of this preparative regimen to facilitate long-term engraftment of allogeneic stem cells and lymphocytes in these patients.
* Determine the response in measurable/evaluable disease and its temporal relationship to the preparative chemotherapy used and to the onset of clinical graft-versus-host disease (GVHD) in patients treated with this regimen.

Secondary

* Determine the progression-free and overall survival of patients treated with this regimen.
* Determine the tumor response and its temporal relationship to administration of high-dose chemotherapy and to the onset of GVHD in patients treated with this regimen.
* Determine the frequency and durability of the induction of full donor chimerism of lymphocytes in patients treated with this regimen.

OUTLINE: This is a nonrandomized, pilot study.

* Nonmyeloablative preparative regimen: Patients receive fludarabine IV over 30 minutes on days -8 to -4, anti-thymocyte globulin IV over 4 hours on days -7 to -4, and high-dose melphalan IV over 30 minutes on days -3 and -2.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV (and then orally when tolerated) every 12 hours beginning on day -4 and tapered after day 42 (if no GVHD occurs) or after day 90 (if grade I acute GVHD occurs). Patients also receive methotrexate IV on days 1, 3, and 6.
* Allogeneic peripheral blood stem cell transplantation (PBSCT): Patients undergo allogeneic PBSCT on day 0. Patients also receive filgrastim (G-CSF) IV or subcutaneously beginning on day 0 and continuing until blood counts recover.
* Donor lymphocyte infusion (DLI): Patients who show disease progression or fail to achieve full donor type T-cell chimerism (at least 90% donor derived T-cells) by the 90-day assessment posttransplantation, and have no evidence of active GVHD may receive DLI. Patients who have unresponsive disease with no active GVHD receive subsequent DLIs every 6-8 weeks.

Patients are followed at 1, 3, 6, 12, 18, 24, 30, and 36 months.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Metastatic disease
* Meets 1 of the following criteria:

  * Chemotherapy-unresponsive disease defined as 1 of the following:

    * Less than a partial response to 2 consecutive chemotherapy regimens that included an anthracycline and a taxane in combination or succession
    * Progression of disease during or within 3 months of completion of a taxane, anthracycline, or platinol-based regimen
  * Histologically confirmed tumor involvement on bone marrow biopsy
* Measurable or evaluable disease* defined as the following:

  * Bidimensionally reproducible measurable mass by physical examination, ultrasonography, radiography, CT scan, or MRI
  * Evaluable lesions apparent on clinical exam, x-ray, CT scan, or MRI which do not fit the criteria for measurability (e.g., ill-defined post-surgical masses or masses assessable in 1 dimension only)

    * Elevation of biological markers (e.g., CA 27.29) is considered evaluable disease NOTE: *Bone lesions or pleural or peritoneal effusion alone are not considered measurable or evaluable disease
* Appropriate candidate for allogeneic stem cell transplantation
* No active CNS metastases
* Available HLA-identical sibling donor

  * 6/6 antigen match
  * Donor CD34 cells at least 2 times 10^6/kg recipient weight
* Hormone receptor status:

  * Estrogen receptor negative or positive

    * Estrogen receptor positive tumors must demonstrate progression on at least 1 hormonal manipulation

PATIENT CHARACTERISTICS:

Age

* 18 to 60

Sex

* Female

Menopausal status

* Not specified

Performance status

* Karnofsky 70-100% OR
* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 1,500/mm^3
* Platelet count at least 30,000/mm^3

Hepatic

* Bilirubin less than 3 times normal*
* AST and ALT less than 3 times normal* NOTE: *Unless abnormality due to malignancy

Renal

* Creatinine no greater than 1.6 mg/dL

Cardiovascular

* LVEF greater than 40% by echocardiography or MUGA
* No myocardial infarction within the past 6 months

Pulmonary

* DLCO greater than 40% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No serious localized or systemic infection
* No hypersensitivity to E. coli-derived products
* No history of non-breast malignant disease within the past 5 years except completely excised nonmelanoma skin cancer or carcinoma in situ of the cervix
* No chronic inflammatory disorder requiring concurrent glucocorticosteroids or other immunosuppressive medication
* No psychological condition or social situation that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* No concurrent glucocorticoids

Radiotherapy

* No prior radiotherapy to an indicator lesion unless the lesion shows evidence of progression after discontinuation of the therapy

Surgery

* Not specified

Other

* No concurrent immunosuppressive medication

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2003-07; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward D. Ball, MD, Principal Investigator — University of California, San Diego
Locations (1):
- Rebecca and John Moores UCSD Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The protocol recruited patients with Metastatic breast cancer for transplant after ATG, high-dose Melphalan and Fludarabine.This was a non-randomized, single arm pilot study. Patients received fludarabine IV days -8 to -4, ATG IV on days -7 to -4 and High dose Melphalan days -3 to -2. This protocol is closed to accrual as of March 2008
Groups:
- Treatment: anti-thymocyte globulin
  filgrastim
  graft-versus-tumor induction therapy
  therapeutic allogeneic lymphocytes
  cyclosporine
  fludarabine phosphate
  melphalan
  methotrexate
  peripheral blood stem cell transplantation
Period: Overall Study
Arm/Group | Treatment
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: This is a pilot study. The original planned target accrual was 15 male or female patients age 18-60 but due to poor enrollment the study was closed to accrual early after 5 patients had been enrolled.
Groups:
- Pilot Study of Allogeneic Transplant for Metastatic Breast Can: anti-thymocyte globulin
  filgrastim
  graft-versus-tumor induction therapy
  therapeutic allogeneic lymphocytes
  cyclosporine
  fludarabine phosphate
  melphalan
  methotrexate
  peripheral blood stem cell transplantation
Arm/Group | Pilot Study of Allogeneic Transplant for Metastatic Breast Can
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 45 [40 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 5 years post transplant
Population: study was closed early due to lack of accrual.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Toxicity
  anti-thymocyte globulin
  filgrastim
  graft-versus-tumor induction therapy
  therapeutic allogeneic lymphocytes
  cyclosporine
  fludarabine phosphate
  melphalan
  methotrexate
  peripheral blood stem cell transplantation
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Number of Participants With Long-term Engraftment of Allogeneic Stem Cells and Lymphocytes
Description: Long-term Engraftment of Allogeneic Stem Cells and Lymphocytes based on cell counts of ANC >1000 for 3 consecutive days and platelet count of >50,000
Time Frame: 30 days post transplant
Population: study was closed early due to lack of accrual.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Patients treated on protocol
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 5

3. Primary Outcome: Number of Participants With Acute and Chronic Graft-versus-host Disease (GVHD)
Time Frame: 100 days post transplant
Population: study was closed early due to lack of accrual.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment: Patients Treated Per Protocol
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 3

4. Secondary Outcome: Progression-free Survival
Description: Progression assessed by CT scan
Time Frame: From date of transplant until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
Population: study was closed early due to lack of accrual.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 5
days | 110 [8 to 180]

5. Secondary Outcome: Overall Survival
Time Frame: 1 year from the time of transplant
Population: study was closed early due to lack of accrual.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 5
days | 279.4 [98 to 373]

6. Secondary Outcome: Response as Measured at 12 Months Post Allografting
Description: response (partial and complete) assessed by CT scan at 12 months post allografting
Time Frame: From date of transplant until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Population: study was closed early due to lack of accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 3

7. Secondary Outcome: Frequency of the Induction of Full Donor Chimerism of Lymphocytes as Measured at 1 Month Post Allografting
Time Frame: 1 month post allografting
Population: study was closed early due to lack of accrual.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: 5 years
Description: AEs and SAEs collected on all Patients
Groups:
- Treatment: The events monitored in the treatment arm of the protocol are listed below:
  incidence of Toxicity
  administration of filgrastim
  Grade of GVHD
  Initiation of graft-versus-tumor induction therapy
  Disease Status
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 3/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=5)
Infection (Infections and infestations) | 5 (5)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Fever (Infections and infestations) | 2 (2)
aGVHD Skin (Skin and subcutaneous tissue disorders) | 2 (2)
aGVHD Gut (Gastrointestinal disorders) | 1 (1)
aGVHD Liver (Hepatobiliary disorders) | 2 (2)
Overall GVHD (Immune system disorders) | 3 (3)
Bilteral Conjunctivitis (Eye disorders) | 1 (1)
ALT Elevation (Hepatobiliary disorders) | 2 (3)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
AST Elevation (Hepatobiliary disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Capillary Leak Syndrome (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Terminated early due to small numbers of subjects enrolled on study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No